CLINICAL TRIAL: NCT06776484
Title: Biological Evolution of Whipple's Disease
Brief Title: Biological Evolution of Whipple's Disease (WHIP)
Acronym: WHIP
Status: Completed | Type: Observational
Sponsor: University Hospital, Brest (Other)
Responsible Party: Sponsor
Other Study IDs: 29BRC24.0315 - WHIP
Record Dates: First submitted 2024-12-18; First posted 2025-01-15 (Actual); Last update posted 2025-01-15 (Actual); Status verified 2024-12

CONDITIONS: Whipple Disease
MeSH Terms: conditions — Whipple Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Whipple's disease (WD), a rare systemic infection by Tropheryma whipplei, lacks research on biological abnormalities pre- and post-treatment. This study explores these abnormalities for their diagnostic and monitoring value.

DETAILED DESCRIPTION:
Whipple's disease (WD) is a rare systemic infection caused by *Tropheryma whipplei*. Despite advancements in diagnosis through PCR and biopsy, there is limited research comparing biological abnormalities before and after treatment. This study aimed to characterize these abnormalities and evaluate their potential for aiding in diagnosis and monitoring.

ELIGIBILITY:
Inclusion Criteria:

* Patients with at least one positive PCR test for Whipple's disease and a retained diagnosis at Brest University Hospital between 2010 and 2024
* Major patient

Exclusion Criteria:

* Minors
* No screening test for Whipple's disease
* Opposition to participation
* Protected patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Retrospective study of patients hospitalised in Brest who tested positive for Whipple's disease between 2010 and 2024
Sampling Method: Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2024-09-01 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Biological changes | 1 day
  Biological changes (inflammation, liver function tests, haematology, lymphocyte subpopulations) in patients diagnosed with classic, localised or reactive Whipple's disease

CONTACTS AND LOCATIONS:
Locations (1):
- Chu Brest, Brest, France

IPD SHARING:
Plan to Share IPD: Yes
All collected data that underlie results in a publication
Supporting Information: Study Protocol
Time Frame: Data will be available beginning three years and ending fifteen years following the final study report completion
Access Criteria: Data access requests will be reviewed by the internal committee of Brest UH. Requestors will be required to sign and complete a data access agreement